CLINICAL TRIAL: NCT06171880
Title: An Open-label, Randomized, Single Administration, Full Replicated Crossover Phase 1 Clinical Trial to Compare Pharmacokinetics and Safety Between JLP-1901 and JC-001 in Healthy Subjects
Brief Title: To Evaluate the Safety and Pharmacokinetic Characteristics After the Administration of JC-001 and JLP-1901
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JP-1901-102
Record Dates: First submitted 2023-11-22; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Healthy Adult
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment(Experimental): JLP-1901 (Experimental): Group I(Peroid I-Comparator[JLP-2008], Peroid II-Treatment[JC-001], Period III-Comparator[JLP-2008], Peroid IV-Treatment[JC-001]), Group II(Peroid I-Treatment[JC-001]Comparator[JLP-2008], Peroid II-Comparator[JLP-2008], Period III-Treatment[JC-001], Peroid IV-Comparator[JLP-2008])
  Interventions: Drug: JLP-1901; Drug: JC-001(active comparator)
- Control(Active Comparator): JC-001 (Active Comparator): Group I(Peroid I-Comparator[JLP-2008], Peroid II-Treatment[JC-001], Period III-Comparator[JLP-2008], Peroid IV-Treatment[JC-001]), Group II(Peroid I-Treatment[JC-001]Comparator[JLP-2008], Peroid II-Comparator[JLP-2008], Period III-Treatment[JC-001], Peroid IV-Comparator[JLP-2008])
  Interventions: Drug: JLP-1901; Drug: JC-001(active comparator)

INTERVENTIONS:
Drug: JLP-1901 — administration of JLP-1901
  Other Names: anti-viral
Drug: JC-001(active comparator) — administration of JC-001(tenofovir)
  Other Names: tenofovir

SUMMARY:
To evaluate the safety and pharmacokinetic characteristics after the administration of JC-001 and JLP-1901

DETAILED DESCRIPTION:
An open-label, randomized, single administration, full replicated crossover phase 1 clinical trial to compare pharmacokinetics and safety between JLP-1901 and JC-001 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults over 19 years of age and under 65 years of age at the time of screening test
2. Those with a body mass index (BMI) of 17.5 kg/m2 or more but less than 30.5 kg/m2 and a body weight of 55 kg or more for men and 45 kg or more for women.
3. Those who do not have congenital or chronic diseases within the past 3 years and have no pathological symptoms or findings as a result of internal medical examination
4. Subjects determined to be suitable as a trial subject as a result of tests performed during screening, such as laboratory tests (hematology test, blood chemistry test, urinalysis, virus/bacteria test, etc.) conducted by the investigator according to the characteristics of the drug, vital signs, and electrocardiogram test.

Exclusion Criteria:

1. Those who have history or evidence of clinically significant blood, kidney, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, liver, mental, nervous or immune diseases (excluding simple dental history such as calculus, impacted teeth, wisdom teeth, etc.)
2. Those whd have a history of gastrointestinal disease (esophageal disease such as achalasia or esophageal stricture, Crohn's disease) or surgery (excluding simple appendectomy, hernia surgery, or tooth extraction surgery) that may affect drug absorption ruler
3. A subject who shows the following values as a result of a laboratory test:

   ☞ ALT or AST > 2 times the upper limit of normal range
4. Those with a history of regular alcohol consumption exceeding 210 g/week within 6 months of screening (1 glass (250 mL) of beer (5%) = 10 g, 1 glass (50 mL) of soju (20%) = 8 g , 1 glass of wine (12%) (125 mL) = 12 g)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
AUC over 24H of JLP-1901 | 24 hours
  AUC over 24H
Cmax of JLP-1901 | 24 hours
  Cmax

CONTACTS AND LOCATIONS:
Locations (1):
- Bundang CHA university global clinical trials center Institutional Review Board, Gyeonggi-do, Bundang-gu, South Korea